CLINICAL TRIAL: NCT01614522
Title: Phase II Open Label Study to Evaluate the Biological Activity of ASLAN001 (ARRY 334543) in Patients With Recurrent/Metastatic Gastric, Gastro-oesophageal Junction, and Oesophageal Carcinoma Whose Tumours Are Epidermal Growth Factor Receptor-2 (HER 2) Amplified or Co-expressing Epidermal Growth Factor Receptor-1 (HER-1) and HER-2.
Brief Title: A Clinical Trial Evaluating the Effect of ASLAN001 in Patients With Recurrent/Metastatic Gastric Cancer Whose Tumors Are Either HER-2 Amplified or Co-expressing HER-1 and HER-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ASLAN001-001
Record Dates: First submitted 2012-05-22; First posted 2012-06-08 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Stomach Neoplasms; Cancer of Stomach; Cancer of the Stomach; Gastric Cancer; Gastric Neoplasms
Keywords: Metastatic gastro-oesophageal carcinoma; Recurrent gastro-oesophageal carcinoma; Gastric cancer; HER-1; HER-2
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HER-2 Amplified (Experimental)
  Interventions: Drug: ASLAN001
- HER-1 & HER-2 Co-expression (Experimental)
  Interventions: Drug: ASLAN001

INTERVENTIONS:
Drug: ASLAN001 — ASLAN001 500mg BID

SUMMARY:
The purpose of this study is to determine whether ASLAN001 has an effect in patients with recurrent or metastatic adenocarcinoma of the stomach, gastrooesophageal junction, or lower third of the oesophagus whose tumours over-express HER-1 and HER-2, or whose tumours are HER-2 gene-amplified.

Maximum of 26 patients will participate in South Korea and the patients will be assigned to either group A or group B according to the results of tests done on tumor tissue obtained by biopsy to determine HER-1 and HER-2 status.

DETAILED DESCRIPTION:
About 1 million new cases of gastric cancer were estimated to have occurred in 2008 (988,000 cases, 7.8% of the total), making it currently the fourth most common malignancy in the world, behind cancers of the lung, breast, and colo-rectum. Gastric cancer is also the second leading cause of cancer-related death in both sexes worldwide with 700,000 deaths occurring annually. The incidence and mortality rates for gastric cancer vary widely in different regions of the world. The incidence has dramatically declined in the United States where it ranks seventh as a cause of cancer- related deaths. In the Asia-Pacific region, the highest incidences of gastric cancer can be found in China, Japan, and Korea, where the age standardized incidence rate (ASR) is greater than 20 per 100,000 populations. Intermediate risk countries (ASR 11-19/100,000 population) include Malaysia, Singapore, and Taiwan, while low-risk countries (ASR < 10/100,000 population) include Australia, New Zealand, India, and Thailand.

Approximately 95% of all malignant gastric neoplasms are adenocarcinomas. One of the most striking epidemiologic observations has been the increasing incidence of adenocarcinomas involving the proximal stomach and distal oesophagus including the oesophagogastric junction. These tumours are thought to have different etiologic factors; gastric body and antral lesions are associated with low acid production and Helicobacter pylori infection, whereas cardiac lesions are not associated with either.

The treatment for advanced and un-resectable disease has remained essentially unchanged for the past 2 decades, with platinum and fluoro-pyridine-based combination chemotherapy being the mainstay of therapy. The molecular biology responsible for carcinogenesis, tumour biology, and response to therapy in gastric cancer are active areas of investigation. Amplification and/or over-expression of epidermal growth factor receptor-2 (HER 2) have been found to promote tumourigenesis and to be involved in the pathogenesis of gastric cancer. Recently, data from randomised studies of trastuzumab (Herceptin®) in patients with HER 2 amplification demonstrated significant improvement in outcome in comparison to chemotherapy alone. Studies on a number other molecularly targeted agents used alone or in combination with chemotherapy have been undertaken, or are ongoing. Translational research, undertaken as part of these studies, demonstrates the great molecular heterogeneity of the disease, with multiple growth factor and survival pathways being implicated.

In view of this, successful therapeutic intervention is likely to require both the identification of molecularly defined subsets of disease, and the evaluation of rationally-selected combinations of targeted agents.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 21 years of age or older at the time written informed consent is obtained.
* Patients with histologically confirmed adenocarcinoma of the stomach, gastro-oesophageal junction or distal oesophagus with inoperable locally-advanced metastatic disease.
* Patients with tumours with immunohistochemical evidence of expression of HER-1 (at level of + or ++ or +++) and HER-2 (at level of + or ++ or +++) using standard criteria OR tumours with gene-amplification of HER-2 by standard FISH.
* Patient has received 1 or more prior chemotherapy for the treatment of adenocarcinoma of the stomach, gastro-oesophageal junction or distal oesophagus with metastatic disease.
* Patients with prior partial gastrectomy if they can take oral medications, and can undergo gastroendoscopic biopsies and meet all other inclusion/exclusion criteria.
* Patients with measurable and non-measurable disease per modified RECIST guidelines. All scans and x-rays used to document measurable or non-measurable disease must be done within a 28-day period prior to enrollment.
* Patient with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (within 14 days prior to enrolment).
* Patient with adequate organ and haematological function as evidenced by the following laboratory studies within 14 days prior to enrollment:
* Haematological function, as follows:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 75 x 109/L
* Haemoglobin ≥ 9 g/dL
* Coagulation functions, as follows:
* Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x upper limits of normal (ULN) per institutional laboratory normal range
* International normalized ratio (INR) ≤ 1.5
* Renal functions, as follows:
* Serum creatinine ≤ 1.5 x ULN
* Urea ≤ 1.5 x ULN
* Hepatic function, as follows:
* Total bilirubin ≤ 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) and serum glutamic pyruvic transaminase (SGPT)/ alanine transaminase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present)*.

  * Except where due to direct disease involvement of the liver at the discretion of the investigator.

Exclusion Criteria:

* Patients unable to swallow oral medications
* Patients with persistent gastric outlet obstruction, complete dysphagia or feeding jejunostomy.
* Patients who underwent radiotherapy to the gastric remnant ≤ 14 days prior to enrolment. Patients must have recovered from all radiotherapy-related toxicities.
* Patients with total gastrectomy.
* Patients who have uncontrolled, clinically significant symptomatic cardiovascular diseases within 6 months prior to enrolment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure or arrhythmias not controlled by outpatient medication.
* Patients with ongoing or clinically significant active infection as judged by the Investigator.
* Pregnant (i.e., positive beta-human chorionic gonadotropin test) or is breast-feeding women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The percentage of patients demonstrating clear evidence of inhibition of receptor auto-phosphorylation in HER-2 amplified patients on Day 29. | Day 29
The percentage of patients demonstrating clear evidence of inhibition of receptor auto-phosphorylation in HER-1 and HER-2 co-expressing patients on Day 29. | Day 29

SECONDARY OUTCOMES:
The percentage of patients showing inhibition of AKT phosphorylation on Day 29. | Day 29
The percentage of patients showing inhibition of MAPK phosphorylation on Day 29. | Day 29
The percentage of patients showing inhibition of Ki67 on Day 29. | Day 29
The percentage of patients showing induction of apoptosis as measured by TUNEL on Day 29. | Day 29
Objective Response Rate | Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, Dr., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Bundang, Seoul
  - Seoul National University Hospital, Seoul